CLINICAL TRIAL: NCT06325969
Title: Evaluation of Immune Status in Patients With Polycystic Ovary Syndrome
Brief Title: PCOS Patients' Immune Alterations
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Prof., Shanghai 10th People's Hospital
Other Study IDs: PCOS Immune
Record Dates: First submitted 2024-03-08; First posted 2024-03-22 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Polycystic Ovary Syndrom; Metformin; Immune Function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women with PCOS: Women aged 18 to 45 who meet the 2003 Rotterdam criteria for PCOS.
  Interventions: Diagnostic Test: Detect the immune function of peripheral blood samples
- Women without PCOS: Non-PCOS women aged 18 to 45.
  Interventions: Diagnostic Test: Detect the immune function of peripheral blood samples

INTERVENTIONS:
Diagnostic Test: Detect the immune function of peripheral blood samples — Flow cytometry was used to detect the immune function of peripheral blood samples of PCOS patients.

SUMMARY:
In this study, the investigators will include PCOS patients and healthy women who meet the trial criteria from the clinical research centers of 3 hospitals, introduce the content of this study to participants, and invite participants to participate. Flow cytometry was used to detect the immune function of peripheral blood samples of PCOS patients, to clarify the immune function characteristics of PCOS patients, and to try to establish an evaluation method of the immune function of PCOS patients.

DETAILED DESCRIPTION:
PCOS patients and healthy women were recruited in outpatient clinics of three hospitals, and peripheral blood was retained for flow cytometry after completing relevant examinations. In this study, flow cytometry was used to detect the antigenic antibody reaction between the surface differentiation antigen of lymphocyte membrane and fluorescence-labeled antibody in human peripheral blood, and the unlabeled cells were dissolved. The number and percentage of cell groups expressing different markers were counted by the fluorescence detection system on flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged 18-45 years;
* Voluntarily participate in the experiment, willing to sign the informed consent.
* According to the Rotterdam consensus, polycystic ovarian syndrome (PCOS) needs to meet the presence of two of three of the following criteria: oligo-anovulation, hyperandrogenism, and polycystic ovaries (≥ 12 follicles measuring 2-9 mm in diameter and/or an ovarian volume > 10 mL in at least one ovary).

Exclusion Criteria:

* Female patients younger than 18 years old or older than 45 years old;
* Ovulation disorders caused by premature ovarian failure, pituitary amenorrhea, hypothalamic amenorrhea, and thyroid dysfunction (hyperthyroidism, hypothyroidism);
* Congenital adrenal hyperplasia, Cushing's syndrome, hyperprolactinemia, adrenal tumors, and other diseases causing hyperandrogenemia;
* Severe liver and kidney dysfunction (more than 3 times the normal value)
* Type 1 diabetes, monogenic mutation diabetes, diabetes due to pancreatic injury or other secondary diabetes;
* History of malignant tumor;
* Severe infection, severe anemia, neutropenia, and other chronic diseases of the system;
* Patients undergoing total hysterectomy or ovarian adnexectomy;
* Mental illness, dementia, or other cognitive behavioral problems;
* Hypoglycemic drugs that may affect insulin resistance and androgen levels, including thiazolidinedione, metformin, SGLT-2i, acarbose, and glucagon-like peptide-1 receptor agonist (GLP-1RA), have been used in the past 3 months;
* Take letrozole, clomiphene, oral contraceptives, glucocorticoids, gonadotropins, gonadotropin-releasing hormone agonists, antiandrogens (spironolactone, cyproterone acetate, flutamide, etc.), and other medications for PCOS treatment within the last 3 months.
* Pregnant or lactating patients;
* Female patients with a BMI less than 20kg/m2.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women older than 18 years or younger than 45 years.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
The number of cell groups expressing different markers were counted by the fluorescence detection system on flow cytometry. | Samples to be collected once per participant within 7 days of enrollment.
  Flow cytometry was used to detect the antigenic antibody reaction between the surface differentiation antigen of lymphocyte membrane and the fluorescently labeled antibody in human peripheral blood, and the unlabeled cells were dissolved.
The percentage of cell groups expressing different markers were counted by the fluorescence detection system on flow cytometry. | Samples to be collected once per participant within 7 days of enrollment.
  Flow cytometry was used to detect the antigenic antibody reaction between the surface differentiation antigen of lymphocyte membrane and the fluorescently labeled antibody in human peripheral blood, and the unlabeled cells were dissolved.

SECONDARY OUTCOMES:
Homeostasis model assessment of insulin resistance | Within 7 days of enrollment.
  insulin resistance index
body mass index | Within 7 days of enrollment.
  body mass index (kg/m2)
menstrual frequency | Within 7 days of enrollment.
  number of menstruation in a year
fasting glucose | Within 7 days of enrollment.
  fasting glucose (mmol/L)
fasting insulin | Within 7 days of enrollment.
  fasting insulin (mmol/L)
Total cholesterol | Within 7 days of enrollment.
  Total cholesterol (mmol/L)
Triglycerides | Within 7 days of enrollment.
  Triglycerides (mmol/L)
HDL-c | Within 7 days of enrollment.
  HDL-c (mmol/L)
LDL-c | Within 7 days of enrollment.
  LDL-c (mmol/L)
total testosterone | Within 7 days of enrollment.
  total testosterone (nmol/L)
free testosterone | Within 7 days of enrollment.
  free testosterone (nmol/L)
Sex hormone-binding globulin | Within 7 days of enrollment.
  Sex hormone-binding globulin (nmol/L)
Androstenedione | Within 7 days of enrollment.
  Androstenedione (ng/ml)
Dehydroepiandrosterone | Within 7 days of enrollment.
  Dehydroepiandrosterone (ug/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Manna Zhang, doctor, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Department of Endocrinology, Shanghai Tenth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No